CLINICAL TRIAL: NCT06070714
Title: Multi-Center Randomized Clinical Trial Evaluating the Efficiency and Safety of Holmium Laser With Moses Technology Versus SuperPulsed Laser System With Thulium Fiber Laser on Renal Stones
Brief Title: Efficiency and Safety of Holmium Laser With Moses Technology Versus SuperPulsed Laser System With Thulium Fiber Laser on Renal Stones
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0932; Urology (Other: UW Madison); Protocol Version 5/21/24 (Other: UW Madison)
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (ratio 1:1) to be treated with either the holmium laser with pulse modulation or the thulium fiber laser. Each site will randomize their own participants. Block randomization in block sizes of 4 will be used to assign participants to each laser treatment group. If unable to use the specified laser for any reason, the participant will be considered a withdrawal
Who Masked: Outcomes Assessor
Masking Description: A single urologist will evaluate all CT scans for residual stones and will be blinded to which laser was used during ureteroscopy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Holmium laser with pulse modulation (Active Comparator)
  Interventions: Device: Holmium laser with pulse modulation
- Thulium fiber laser (Active Comparator)
  Interventions: Device: Thulium fiber laser

INTERVENTIONS:
Device: Holmium laser with pulse modulation — The holmium laser with pulse modulation emits two separate laser pulses with a short time interval between them. The first pulse divides the water between the laser fiber tip and the stone and the second pulse hits the stone unobstructed.
  Arms: Holmium laser with pulse modulation
Device: Thulium fiber laser — The thulium fiber laser has a different wavelength then the holmium laser with pulse modulation and thus has slightly different energy properties. It has also been shown to increase ablative volume and decrease retropulsion without any safety concerns.
  Arms: Thulium fiber laser

SUMMARY:
This is a prospective randomized controlled trial designed to assess the efficacy and safety of Lumenis® Pulse™ P120H holmium laser system with the Moses technology (holmium laser with pulse modulation) versus the Soltive™ SuperPulsed Laser System with the thulium fiber laser (thulium fiber laser), in dusting of renal stones during ureteroscopy with laser lithotripsy. 310 participants will be enrolled across 5 research sites.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial comparing ureteroscopy with laser lithotripsy with the Lumenis® Pulse™ P120H holmium laser system with the Moses technology (holmium laser with pulse modulation) versus the Soltive™ SuperPulsed Laser System with the thulium fiber laser technology (thulium fiber laser).

The primary objective is to compare the stone free rate as determined by computed tomography (CT) scan at two months (6-10 weeks) post operatively. A single urologist will evaluate all CT scans for residual stones and will be blinded to which laser was used during ureteroscopy.

The following information will be collected for research purposes as secondary outcomes: (1) stone treatment time (time from the start of lasing to the end of lasing; minutes); (2) total operative time (minutes); (3) lasing time (minutes, time the laser was in use, not including pedal pauses); (4) total energy used (kilojoules, kJ); (5) laser efficiency (mm per minute); (6) number of times the laser pedals are pressed (left, right, and total pedal presses); (7) laser fiber size; (8) stone analysis; (9) complications, and (10) patients' quality of life.

The results from the pre- and post-operative quality of life survey (WISQOL short form) will be obtained from the patient's medical record. A total of 3 clinic visits (i.e., the pre-operative visit and the stone surgery, one post-operative visit after 2 months of the surgery) will be needed for this study.

All visits are standard of care. Stone parameters (i.e. size, location, Hounsfield units, presence of hydronephrosis, stone volume, and composition), demographic information, co-morbidities, and post-operative parameters will be collected from the medical record in HealthLink.

The Thulium laser company is not involved in this research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal stones who require endoscopic laser treatment in the outpatient operating room. Patients may have an ureteropelvic junction (UPJ) stone if the treatment of the stone is completed in the kidney.
* Patients' stone size in a single renal unit of greater than or equal to 5 millimeters (mm) and less than or equal to 20 mm. Stone size is defined as the largest diameter of a single stone on pre-operative CT as assessed by the urologist. Patients with multiple stones will be included as long as their largest stone size falls within the above parameters.

Exclusion Criteria:

* Pregnant patients
* Patients with transplant kidneys or other anatomic variations: horseshoe kidney, pelvic kidney, ptotic kidney, urinary diversion or ureteral stricture
* Patients with irreversible coagulopathy
* Patients with known ureteral stricture disease
* Patient who do not have a pre-operative CT
* Non-English speaking patients and patients in other vulnerable groups such as lacking of decision-making capability, prisoner, or adult unable to consent
* Uric acid composition greater than 50 percent on pre operative stone analysis. Patients will be excluded post operatively if stone analysis from the time of surgery is greater than 50 percent uric acid.
* Prior ureteroscopy within 6 weeks of current surgery
* Urothelial tumor(s), direct extraction of the stone(s) without needing laser lithotripsy, and failure to reach the stone in the upper urinary tract with the ureteroscope
* Patients with only ureteral stones (ureteropelvic junction stones may be included as long as treated in the kidney)
* Patients with renal tubular acidosis or medullary sponge kidney

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Stone Free Rate | 2 months post-op (up to 10 weeks on study)
  The primary objective of this study is to compare the stone free rate as determined by ultra-low dose limited renal CT at 2 months post operatively between the holmium laser with pulse modulation and the thulium fiber laser.

SECONDARY OUTCOMES:
Stone Treatment Time in Minutes | day of procedure (up to 3 hours)
  Time from the start of lasing to the end of lasing.
Total Operative Time in Minutes | day of procedure (up to 3 hours)
Procedural time | day of procedure (up to 3 hours)
  time from the insert to removal of the instrument
Total Energy Used in kilojoules | day of procedure (up to 3 hours)
Laser Efficiency in millimeters per minute | day of procedure (up to 3 hours)
Number of Participants with Procedural Complications | day of procedure (up to 3 hours)
Participant Quality of Life as Measured by the WISQOL Short Form Score | pre-operative (baseline) and post-operative (up to 10 weeks)
  WISQOL short form is a 6 item questionnaire which can be scored from 1(worst outcome) to 5 (best outcome). The raw score range is 5-30. In the study, standardized total score is used. the range of the standardized total score is 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nakada, MD, FACS, FRCS, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - University of California - Los Angeles, Los Angeles, California
  - Mount Sinai Health System, New York, New York
  - Glickman Urological & Kidney Institute, Cleveland, Ohio
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No